CLINICAL TRIAL: NCT01289652
Title: PRospective OBservational Evaluation of the Natural History and Treatment of Acute HCV in HIV-positive Individuals: The PROBE-C Study
Brief Title: The Natural History and Treatment of Acute Hepatitis C Virus (HCV) in HIV-positive Individuals
Acronym: PROBE-C
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Benedetta Mattioli (Other)
Responsible Party: Sponsor-Investigator, Benedetta Mattioli, MD, Istituto Superiore di Sanità
Organization: Istituto Superiore di Sanità (Other)
Other Study IDs: PROBE-C V 2.3, 03 June 20; NEAT (Other Grant/Funding Number: NEAT002)
Record Dates: First submitted 2011-02-03; First posted 2011-02-04 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Acute Hepatitis C; HIV
Keywords: Acute hepatitis C (HCV); Human immunodeficiency virus (HIV)
MeSH Terms: conditions — Hepatitis C; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For phylogenetic analysis HCV RNA detection will be performed.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- HCV + HIV
- HCV

SUMMARY:
The aim of the study is to investigate the epidemiology, natural history and treatment outcomes of acute hepatitis C (HCV) infection. Given the current pattern of case reporting, the cohort will be largely made up of human immunodeficiency virus (HIV)-positive patients, but HIV-negative patients with acute hepatitis C (AHC) will also be enrolled to enable comparisons to be made as appropriate and possible.

DETAILED DESCRIPTION:
In a multi-center, prospective, open cohort study, patients with documented acute hepatitis C infection will be followed prospectively over an initial time-period of 3 years after diagnosis of acute hepatitis C infection to investigate:

1. epidemiology

   * to describe the characteristics of patients who have acquired acute HCV infection, including examination of regional differences in modes of transmission, behavioural factors, concomitant sexually transmitted diseases, clinical presentation and associated laboratory test results.
   * characterization of the HCV strains circulating within the community using phylogenetic analysis
2. natural history

   * determination of the rate of spontaneous viral clearance, and the clinical, immunological, host genetic and viral factors associated with viral clearance
   * progression of liver disease after acute hepatitis C; including the use of non-invasive liver fibrosis markers to estimate rates of liver fibrosis progression
3. treatment strategies

   * describe the outcome of different treatment strategies for acute HCV infection, although it is acknowledged that there will be no random allocation of treatment strategies.
   * investigate factors associated with treatment response including time to initiation of therapy, duration of therapy, the use of ribavirin and genetic factors.

ELIGIBILITY:
Inclusion Criteria:

* Documented current or past acute hepatitis C infection with detectable HCV-RNA (PCR-assay) with an estimated duration of 52 weeks at diagnosis as defined below:

  * First HCV RNA positive AND
  * Prior negative anti-HCV antibody or HCV RNA test within 12 months OR
  * Rise of liver transaminases above 2.5 x upper limit of normal (ULN) within the past 12 months with prior normal transaminases during the year before AND
  * Exclusion of other causes of acute hepatitis

Exclusion Criteria:

* Acute liver disease other than hepatitis C
* Inability to provide written informed consent
* Younger than 18 years of age

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 600 acute HCV infections with/without HIV infection
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2011-05; Primary Completion 2016-05 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
SVR | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Bonn University Hospital, Bonn, NSW, Germany